CLINICAL TRIAL: NCT02070419
Title: Trans-Arterial Chemo-Embolization (TACE) vs TACE Plus Stereotactic Body Radio Therapy (SBRT) in the Treatment of Hepatocellular Carcinoma (HCC)
Brief Title: TACE With or Without Radiation Therapy in Treating Patients With Stage A-C Liver Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE2212; NCI-2014-00246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE2212; CASE 2212 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Recurrent Adult Primary Liver Cancer; Stage I Adult Primary Liver Cancer; Stage II Adult Primary Liver Cancer; Stage IIIA Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (TACE) (Active Comparator): Patients undergo (transarterial chemoembolization) TACE according to institutional standard with doxorubicin-eluting beads.
  Interventions: Procedure: transarterial chemoembolization
- Arm II (TACE+SBRT) (Experimental): Patients undergo transarterial chemoembolization (TACE) as in Arm I and 3 or 5 fractions of stereotactic radiosurgery (SBRT) given at least 48 hours apart over 14 days.
  Interventions: Procedure: transarterial chemoembolization; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Procedure: transarterial chemoembolization — Undergo TACE with doxorubicin-eluting beads
  Other Names: TACE
Radiation: stereotactic radiosurgery — Undergo SBRT
  Arms: Arm II (TACE+SBRT)

SUMMARY:
This randomized phase II trial studies how well transarterial chemoembolization (TACE) works compared with TACE plus radiation therapy in treating patients with end stage liver disease, liver tumors, or potential liver transplant candidates. TACE involves reaching up to the blood vessel that feeds the tumor through a catheter placed into the groin vessel. Once the physician has defined the vessel going to the tumor, chemotherapy is infused to the tumor and the vessel is blocked, maintaining the chemotherapy for longer time inside the tumor and stopping the blood flow that feeds the tumor. Stereotactic body radiation therapy (SBRT) is a type of radiation therapy that delivers radiation to the tumor cells but does not harm normal liver cells. It is not yet known whether TACE is more effective with or without SBRT in treating liver tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine in patients with stage A to C hepatocellular carcinoma, if stereotactic body radiotherapy after TACE enhanced the response rate of hepatocellular carcinoma (HCC) when compared to TACE alone at 3 months.

SECONDARY OBJECTIVES:

I. To determine in patients with stage A to C hepatocellular carcinoma, if TACE plus SBRT can achieve a downstaging rate of >= 30% at 3 and 6 months.

II. To determine the rate of grade 3 or 4 adverse events associated with SBRT for liver tumors.

III. To determine the rate of local progression after SBRT. (Based on Response Evaluation Criteria in Solid Tumors [RECIST] criteria) IV. Number of patients who achieve liver transplantation. V. Overall survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms after the first loco-regional therapy with TACE.

ARM I: Patients undergo TACE according to institutional standard with doxorubicin-eluting beads.

ARM II: Patients undergo TACE as in Arm I and 3 or 5 fractions of SBRT given at least 48 hours apart over 14 days.

After completion of study treatment, patients are followed up at 1, 3, and 6 months and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* HCC is staged as Barcelona A to C
* Treatment with SBRT can occur within 6 weeks of registration
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patient has

  * Radiographic enhancing liver lesions with early wash out on triple phase CT or MRI or
  * Histological confirmation of HCC as determined by the Liver Tumor Board
* Hemoglobin greater than 10.0 g/dL
* Total bilirubin less than 3.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3 X institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal
* Total aggregate of maximal dimension of liver tumors is =< 8 cm
* Cirrhotic patients Child Pugh class A or B (score =< 7)
* Patient must be determined by the treating physician to be medically eligible for liver transplantation measured by imaging modality (magnetic resonance imaging [MRI]/computed tomography [CT] scan) three months post final treatment
* Absolute neutrophil count >= 1,500/μl
* Platelet count >= 50,000 μl (after transfusion if required)
* Life expectancy > 12 weeks
* Subjects must have the ability to understand and be willing to provide written informed consent
* Women of child-bearing potential must have a negative pregnancy test within 4 weeks to the start of the SBRT treatment
* Women must not be pregnant or nursing
* Sexually active women must agree to use accepted forms of birth control; acceptable options for birth control will be documented in the consent and discussed with the subject prior to enrollment

Exclusion Criteria:

* Patient with previous history of abdominal radiation
* Cirrhotic patients Child Pugh class B with score >= 8
* Prior invasive malignancy other than primary liver malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Evidence of metastatic disease prior to registration
* Evidence of main portal vein thrombosis
* History of known cardiac ischemia or stroke within last 6 months
* Any concurrent medical or psychosocial condition that prohibits a major surgical procedure or immunosuppression that would constitute a contraindication to liver transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage change in gross tumor volume (GTV) | Baseline to 3 months
  Percentage of tumor response as defined as change in longest diameter of tumor compared to original tumor length
Difference in mean gross tumor volume (GTV), assessed using the RECIST method | Baseline to 3 months
  Difference in mean GTV from T0M and T3M calculated by a student t-test
Difference in tumor grade | Baseline to 3 months
  Difference in the grade of tumor (as defined by the RECIST criteria) at T0 and T3 calculated using Chi-square tests.

SECONDARY OUTCOMES:
Rate of downstaging | Up to 6 months
  Rate of downstaging of stage A to C Hepatocellular Carcinoma using TACE plus SBRT when compared to TACE at 3 and 6 months.
Grade 3 or 4 adverse events associated with liver tumors | Up to 1 year
  Number of grade 3 or 4 adverse events associated with SBRT for liver tumors, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events
Rate of local progression, based on RECIST criteria | Up to 6 months
  Rate of local disease progression when progression is defined as an estimated increase of > 20% in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Liver transplant achievement | Up to 6 months
  Number of patients who achieve liver transplantation
Survival rate | 1 year
  The number of days from the first day of treatment on study until death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanabria, Principal Investigator — Case Comprehensive Cancer Center